CLINICAL TRIAL: NCT00385593
Title: A Comparison of Symbicort Single Inhaler Therapy (Symbicort Turbuhaler 160/4.5 Micrograms, 1 Inhalation b.i.d. Plus as Needed) and Conventional Best Practice for the Treatment of Persistent Asthma in Adults - a 26-week, Randomised, Open-label, Parallel-group, Multicentre Study. Study SPAIN
Brief Title: Symbicort Single Inhaler Therapy vs Conventional Best Practice for the Treatment of Persistent Asthma in Adults
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D5890L00010; 2005-005974-64; SPAIN
Record Dates: First submitted 2006-10-06; First posted 2006-10-09 (Estimated); Results first posted 2009-11-17 (Estimated); Last update posted 2010-12-16 (Estimated); Status verified 2010-11

CONDITIONS: Asthma, Bronchial
MeSH Terms: conditions — Asthma | interventions — Budesonide, Formoterol Fumarate Drug Combination; Budesonide; Formoterol Fumarate

INTERVENTIONS:
Drug: Symbicort (budesonide/formoterol) Turbuhaler
Drug: Conventional treatment

SUMMARY:
This study is intended to extend the knowledge of Symbicort Single Inhaler Therapy into a more general setting in order to assess the real-life impact of introducing this new treatment concept. The study will compare the Symbicort Single Inhaler Therapy concept with a conventional stepwise treatment regimen according to the investigator's judgement in patients who present with symptoms on inhaled glucocorticosteroids (GCS) treatment or who require and are already on treatment with a combination of inhaled and long-acting B2 agonists (LABA).

ELIGIBILITY:
Inclusion Criteria:

* Minimum of 3 months history of asthma, diagnosed according to the American Thoracic Society (ATS) definition (9).
* Prescribed inhaled GCS at a dose of 400μg/day of budesonide (or equivalents)and within the approved label for the relevant drug during the last 3 months prior to Visit 1.
* Either daily maintenance treatment with both inhaled GCS and LABA or daily treatment with inhaled GCS alone (i.e. without LABA)
* A history of suboptimal asthma control the month prior to enrolment as judged by the investigator
* Use of ≥3 inhalations of as needed medication for symptom relief during the last 7 days before enrolment

Exclusion Criteria:

* Previous treatment with Symbicort Single Inhaler;
* Use of any b-blocking agent, including eye-drops and oral GCS as maintenance treatment.
* Known or suspected hypersensitivity to study therapy or excipients.
* A history of smoking ≥ 10 pack years.
* Asthma exacerbation requiring change in asthma treatment during the last 14 days prior to or at Visit 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 654 (Actual)
Dates: Start 2006-09; Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Barcina, MD, Study Director — AstraZeneca
Locations (52):
- Spain (52):
  - Research Site, A Coruña
  - Research Site, Alagón
  - Research Site, Alicante
  - Research Site, Almoradí
  - Research Site, Barcelona
  - Research Site, Burgos
  - Research Site, Cadiz
  - Research Site, Caravaca
  - Research Site, Cartagena
  - Research Site, Coslada
  - Research Site, Córdoba
  - Research Site, Donostia / San Sebastian
  - Research Site, Dos Hermanas
  - Research Site, Elche
  - Research Site, Fuencarral
  - Research Site, Fuenlabrada
  - Research Site, Galdakao
  - Research Site, Gallur
  - Research Site, Gandia
  - Research Site, Getafe
  - Research Site, Gijón
  - Research Site, Granada
  - Research Site, Huelva
  - Research Site, Huesca
  - Research Site, Idiazabal
  - Research Site, Jaén
  - Research Site, Lugo
  - Research Site, Madrid
  - Research Site, Mataró
  - Research Site, Málaga
  - Research Site, Oviedo
  - Research Site, Pamplona
  - Research Site, Pinto
  - Research Site, Pozuelo de Alarcón
  - Research Site, Sagunto
  - Research Site, Salamanca
  - Research Site, San Juan
  - Research Site, Santander
  - Research Site, Santiago
  - Research Site, Santiago de Compostela
  - Research Site, Seville
  - Research Site, Terrassa
  - Research Site, Valdemoro
  - Research Site, Valencia
  - Research Site, Valladolid
  - Research Site, Vigo
  - Research Site, Viladecans
  - Research Site, Vilanova
  - Research Site, Villabona
  - Research Site, Villanueva de la Cañada
  - Research Site, Vitoria-Gasteiz
  - Research Site, Zaragoza

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 654
Groups:
- SMART: Symbicort Turbuhaler 160/4.5μg, 1 inhalation b.i.d. + as needed (in response to symptoms)
- Conv. Best Practice: Conventional best practice, active stepwise individualized treatment according to international asthma treatment guidelines (GINA guidelines)); stepwise treatment according to the investigator's clinical judgement.
Period: Overall Study
Arm/Group | SMART | Conv. Best Practice
Started | 328 | 326
Completed | 270 | 289
Not Completed | 58 | 37
Not completed — Adverse Event | 3 | 2
Not completed — Withdrawal by Subject | 17 | 7
Not completed — Lost to Follow-up | 12 | 8
Not completed — Protocol Violation | 7 | 4
Not completed — Several reasons | 17 | 15
Not completed — Incorrect inclusion | 2 | 0
Not completed — Incorrect randomization | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SMART | Conv. Best Practice | Total
Number analyzed (Participants) | 328 | 326 | 654
Age Continuous [Mean (Standard Deviation); unit: Years] | 43.7 (16.4) | 44.3 (16.5) | 44.0 (16.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 218 | 202 | 420
  Male | 110 | 124 | 234

OUTCOME MEASURES:

1. Primary Outcome: Time to First Severe Asthma Exacerbation
Description: Severe asthma exacerbation is defined as deterioration in asthma leading to at least one of Hospitalization/Emergency room (or equivalent) treatment due to asthma or Oral Glucocorticosteroids (GCS) treatment for at least 3 days.
Time Frame: Baseline up to 6 months
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | SMART | Conv. Best Practice
Number analyzed (Participants) | 328 | 326
Days | 174.39 (1.76) | 178.97 (1.86)

2. Secondary Outcome: Total Number of Severe Exacerbations
Description: Severe asthma exacerbation is defined as deterioration in asthma leading to at least one of Hospitalization/Emergency room (or equivalent) treatment due to asthma or Oral (GCS) treatment for at least 3 days.
Time Frame: Baseline up to 6 months
Measure: Number; unit: Exacerbations
Arm/Group | SMART | Conv. Best Practice
Number analyzed (Participants) | 328 | 326
Exacerbations | 24 | 34

3. Secondary Outcome: Mean Use of as Needed Medication
Description: Mean use of as needed medication during the treatment period
Time Frame: Baseline up to 6 months
Measure: Mean (Full Range); unit: Inhalations
Arm/Group | SMART | Conv. Best Practice
Number analyzed (Participants) | 308 | 320
Inhalations | 1.03 (0) [0 to 6] | 1.02 (0) [0 to 9]

4. Secondary Outcome: Use of Inhaled Steroids
Description: Mean micrograms/day of inhaled steroids (beclomethasone dipropionate equivalents)
Time Frame: Baseline up to 6 months
Measure: Mean (Full Range); unit: micrograms
Arm/Group | SMART | Conv. Best Practice
Number analyzed (Participants) | 328 | 326
micrograms | 799 (250) [250 to 2000] | 1184 (200) [200 to 4000]

5. Secondary Outcome: Change in the Asthma Control Questionnaire(ACQ) Score
Description: The ACQ is a 7-point scale with scores ranging from 0 (very well controlled) to 6 (very badly controlled)
Time Frame: Daily 14 days prior to each of visit 2-4
Measure: Mean (Full Range); unit: Scores on a scale
Arm/Group | SMART | Conv. Best Practice
Number analyzed (Participants) | 301 | 306
Scores on a scale | 0.99 (0.0) [0 to 4] | 1.08 (0.0) [0 to 3.4]

6. Secondary Outcome: Peak Expiratory Flow (PEF)
Description: Peak expiratory flow (PEF)
Time Frame: 6 months (end of the study)
Measure: Mean (Full Range); unit: L/min
Arm/Group | SMART | Conv. Best Practice
Number analyzed (Participants) | 285 | 299
L/min | 405.9 [110 to 900] | 400.6 [140 to 900]

ADVERSE EVENTS:
Description: The safety analysis set included 652 patients, because two patients in the Symbicort SMART arm were excluded from the safety analysis because they didn't take any dose of medication
Arm/Group | SMART | Conv. Best Practice
Serious Adverse Events (participants affected / at risk) | 10/326 | 5/326
Other Adverse Events (participants affected / at risk) | 0/326 | 0/326
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SMART (N=326) | Conv. Best Practice (N=326)
Gastroenteritis (Gastrointestinal disorders) | 1 | 0
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Epicondylitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Gene Mutation (Congenital, familial and genetic disorders) | 1 | 0
Medullary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Irritable Bowel Syndrome (Gastrointestinal disorders) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Respiratory Tract Infection (Infections and infestations) | 1 | 0
Cataract (Eye disorders) | 1 | 0
Cerebral Haemorrhage (Vascular disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Bursitis Infective (Infections and infestations) | 0 | 1
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1

LIMITATIONS AND CAVEATS:
The study was prematurely stopped, because it was not possible to recruit the sample size required in the period of time established.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No